CLINICAL TRIAL: NCT06966440
Title: Assessing the Impact of Ct-DNA MRD-Guided Adjuvant Therapy on Outcomes in Resectable Pancreatic Cancer
Brief Title: Adjuvant Pancreatic Therapy Guided by MRD
Acronym: ADAPT-MRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, BAIYONG SHEN, Chief Physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-C2504015-PC
Record Dates: First submitted 2025-04-21; First posted 2025-05-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Adenocarcinoma Resectable

STUDY DESIGN:
Masking Description: The adjuvant chemotherapy regimens in this study include, but are not limited to: GEM monotherapy/adjustable GEM monotherapy, S-1 monotherapy/adjustable S-1 monotherapy, fluorouracil monotherapy/adjustable fluorouracil monotherapy, GEM plus CAP regimen/adjustable GEM plus CAP regimen, mFOLFIRINOX regimen, GEM plus nab-paclitaxel regimen/adjustable GEM plus nab-paclitaxel regimen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: MRD-guided adjuvant treatment (Experimental): In the experimental group, patients will receive a guideline-recommended adjuvant therapy regimen chosen by their physician, with each treatment cycle lasting 12 weeks. MRD testing will be performed before the start of the first treatment cycle, and at weeks 8 and 11 after the start of treatment. If two consecutive MRD tests after the start of treatment are negative, treatment will be discontinued, and the patient will undergo regular follow-up only. Otherwise, another treatment cycle will be added. Starting from the second cycle, MRD testing will only be performed at weeks 8 and 11 of each cycle. If two consecutive MRD tests are negative, treatment will be discontinued, and the patient will undergo regular follow-up (every 8 weeks). Otherwise, treatment cycles will continue until disease progression, patient intolerance to treatment, or study termination.
  Interventions: Diagnostic Test: circulating tumor DNA (ctDNA)-based MRD; Drug: adjuvant chemotherapy regimens
- Arm B: non-MRD-driven, standard of care adjuvant treatment (Placebo Comparator): The control group will receive standard post-operative adjuvant therapy (according to CSCO guideline-recommended treatment duration, generally 6 months) followed by regular follow-up (every 8 weeks).
  Interventions: Drug: adjuvant chemotherapy regimens

INTERVENTIONS:
Diagnostic Test: circulating tumor DNA (ctDNA)-based MRD — MRD testing will be performed before the start of the first treatment cycle, and at weeks 8 and 11 of each subsequent cycle. MinerVa Prime is a tumor-informed MRD assay based on a fixed panel spanning 769 cancer-related genes.
  Other Names: MinerVa
  Arms: Arm A: MRD-guided adjuvant treatment
Drug: adjuvant chemotherapy regimens — Patients will be administered with appropriate adjuvant chemotherapy regimens including but are not limited to: GEM monotherapy/adjustable GEM monotherapy, S-1 monotherapy/adjustable S-1 monotherapy, fluorouracil monotherapy/adjustable fluorouracil monotherapy, GEM plus CAP regimen/adjustable GEM plus CAP regimen, mFOLFIRINOX regimen, GEM plus nab-paclitaxel regimen/adjustable GEM plus nab-paclitaxel regimen.

SUMMARY:
Pancreatic adenocarcinoma (PAAD) is a leading cause of cancer-related deaths worldwide. Although surgical resection can be curative, the 5-year overall survival (OS) rate after resection alone is approximately 20%. Adjuvant chemotherapy can improve survival outcomes in patients with resected PAAD. This study will explore the application of ctDNA MRD in guiding adjuvant therapy in these patients.

This prospective, randomized, interventional trial will evaluate a ct-DNA MRD-guided adjuvant therapy strategy in PAAD patients who have undergone radical resection at our institution. Prior to adjuvant chemotherapy, patients will be randomized (1:1) to either the experimental arm (Arm A) or the control arm (Arm B). Arm A will receive ct-DNA MRD-guided therapy, while Arm B will receive non-ctDNA-driven standard of care post-operative adjuvant therapy.

In Arm A, patients will receive a physician-selected, guideline-recommended adjuvant therapy regimen in 12-week cycles. ctDNA MRD will be assessed before the end of first cycle and at weeks 8 and 11. If two consecutive post-treatment MRD tests are negative, therapy will be "de-escalated" (discontinued) with regular follow-up as determined by the clinician. Otherwise, another treatment cycle will be administered, with the same MRD assessment. Following the second cycle, patients without two negative MRD results (only tested at week 8 and week 11 within each cycle) will "escalate" to a longer duration of chemotherapy (comparing to the 6-month standard of care) at the clinician's discretion. Treatment will continue until disease progression, intolerance, or study termination.

Arm B will receive standard post-operative adjuvant therapy for a duration recommended by CSCO guidelines (typically 6 months), followed by regular follow-up every 8 weeks.

The primary endpoint is to compare the prognosis, tolerability, and treatment completion rates between the two arms.

DETAILED DESCRIPTION:
In pancreatic cancer, circulating tumor DNA (ctDNA) carries tumor-specific mutations (e.g., KRAS, TP53), which can be tracked using next-generation sequencing (NGS) technology to detect minimal residual disease (MRD) after surgery. Previous observational studies suggest that ctDNA-positive patients have a significantly higher risk of postoperative recurrence. In the MRD window (2-12 weeks post-surgery), the median disease-free survival (DFS) for ctDNA-positive patients was only 6.37 months, compared to 33.31 months for ctDNA-negative patients (HR=5.45), indicating that ctDNA-positive patients may require intensified treatment. Furthermore, patients with persistent ctDNA positivity after completing adjuvant chemotherapy (e.g., gemcitabine) still have a high recurrence rate (70%-90%), suggesting the need for alternative treatment strategies.

In a previous study (NCT05479708) evaluating postoperative MRD detection using plasma ctDNA to assess survival benefits and optimize adjuvant chemotherapy strategies in resectable pancreatic cancer patients, we found that MRD-positive patients at 4-8 weeks post-surgery (Landmark MRD) had a higher risk of recurrence. Analysis from Landmark MRD to 36 weeks post-treatment showed that patients who converted from positive to negative MRD status (MRD clearance) had a significantly lower risk of recurrence compared to those who remained positive and those who converted from negative to positive, and MRD clearance was associated with significantly improved overall survival (OS).

Given the significant trauma of pancreatic surgery and the often poor postoperative physical condition of patients, the optimal adjuvant chemotherapy regimen (single-agent/combination, duration, initiation time, etc.) that balances patient recovery and recurrence control remains unclear. Serum biomarker CA 19-9 is commonly used to assess prognosis in pancreatic cancer but is not a reliable predictor of adjuvant therapy efficacy. Imaging methods such as CT/MRI are often used to assess residual tumor or recurrence risk, but their sensitivity and specificity are limited, making it difficult to accurately evaluate real-time tumor burden. Therefore, we designed a prospective, randomized, interventional clinical trial based on ctDNA MRD to guide adjuvant chemotherapy decisions in patients with radically resected pancreatic cancer. The aim is to evaluate whether a ctDNA-guided treatment approach can reduce the use of adjuvant chemotherapy in low-risk patients without increasing recurrence risk, while intensifying treatment in high-risk patients to improve prognosis.

A ctDNA MRD-guided adjuvant therapy approach can allow patients to receive individualized adjuvant treatment. When ctDNA MRD test results are negative, adjuvant chemotherapy can be stopped with active follow-up. This can ensure that clinical benefits are not compromised while avoiding unnecessary chemotherapy. In cases where ctDNA MRD remains positive, continuing treatment can provide patients with more intensive therapy and potentially lead to better prognoses.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing written informed consent (ICF) and able to understand and agree to comply with the study requirements and assessment schedule
* Male or female aged 18-75 years at the time of ICF signing.
* Histologically confirmed pancreatic ductal adenocarcinoma, Stage I-III, and has undergone R0 resection.
* Time between surgery and randomization ≤ 12 weeks.
* ECOG PS 0-2.
* Fully recovered from surgery and able to receive adjuvant chemotherapy.
* Availability of sufficient tumor tissue for MRD testing.
* Patients with reproductive potential (female patients: must have entered the study after the menstrual period and with a negative pregnancy test) must agree to use two medically acceptable methods of contraception (one used by the patient and one by their partner) during the study and for 4 months (for females) or 6 months (for males) after the last study treatment.

Exclusion Criteria:

* Other types of non-ductal pancreatic tumors, including neuroendocrine tumors or acinar cell carcinoma, cystadenocarcinoma, and ampullary carcinoma.
* Hepatic or renal dysfunction as follows, or if the investigator considers adjuvant chemotherapy to be clearly contraindicated: a) Moderate/severe renal impairment (GFR < 30 ml/min) calculated using the Cockcroft-Gault equation. b) Absolute neutrophil count < 1.5 × 10^9/L. c) Platelet count < 100 × 10^9/L. d) Hemoglobin < 90 g/L. e) Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) > 2.5 × the upper limit of normal.
* Pregnant or breastfeeding women.
* Any serious or uncontrolled systemic disease, including uncontrolled hypertension, active bleeding, active infection (including hepatitis B, hepatitis C, HIV, etc.), which the investigator deems unsuitable for participation in the study or likely to affect compliance with the study protocol.
* Concurrent presence of another malignancy or a history of malignancy (except for adequately treated carcinoma in situ of the cervix, basal cell carcinoma, or squamous cell carcinoma of the skin)
* Other conditions that the investigator deems unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From the time of randomization up to three years
  To evaluate the impact of ct-DNA MRD-guided adjuvant therapy on disease-free survival (DFS), defined as the proportion of patients alive without objectively documented disease progression from the time of randomization until the 36th month.

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of randomization until the 36th month (3-year OS rate) or until the 60th month(5-years OS rate)
  To evaluate the impact of ct-DNA MRD-guided adjuvant therapy on overall survival (OS), defined as the proportion of patients alive from the time of randomization until the 36th month (3-year OS rate) or until the 60th month(5-years OS rate).
Adjuvant chemotherapy completion rate | From the time of randomization to the end of treatment (arm A: 12 weeks, 24 weeks, 36 weeks, or 48 weeks; arm B: 24 weeks)
  Adjuvant chemotherapy completion rate, defined in the experimental group (arm A) as the proportion of patients completing 1-cycle, 2-cycle, 3-cycle, or 4-cycle treatment based on MRD results (each cycle is about 12 weeks), and in the control group (arm B) as the proportion of patients completing the prescribed chemotherapy duration (generally 2-cycle treatment, about 24 weeks).
Adverse events (AE) and serious adverse events (SAE) rates | From the time of randomization until the date of first recorded adverse events or serious adverse events as mentioned above, assessed up to 60 months (5-years)
  Incidence of AE and SAE assessed via NCI CTCAE version 5.0 in the two treatment modalities.
  Definition of AE Possible adverse events include: drug-related peripheral sensory neuropathy, diarrhea, neutropenia, thrombocytopenia, nausea, vomiting, mucositis, fatigue, and hand-foot syndrome; as well as puncture site infections related to blood draws during the trial.
  Definition of SAE
  Possible serious adverse events include:
  1. Death of the patient;
  2. Life-threatening adverse events, such as Grade 4 non-hematologic toxicity or Grade 4 hematologic toxicity accompanied by fever and bleeding;
  3. Any adverse event requiring hospitalization or prolongation of existing hospitalization;
  4. Irreversible adverse events;
  5. Unexpected adverse events not listed in the drug label that may impact the continuation of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijing Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia L, Pu Q, Kang R, Mei J, Li L, Yang Y, Deng S, Feng G, Deng Y, Gan F, Lin Y, Ma L, Lin F, Yuan Y, Hu Y, Guo C, Liao H, Liu C, Zhu Y, Wang W, Liu Z, Xu Y, Li K, Li C, Chen W, Li Q, Du B, Zhang X, Kou Y, Wang Y, Wu Z, Che G, Chen Y, Shen S, Chen L, Xie D, Liu L. Dynamic ctDNA informs whole-course postoperative precise management of NSCLC (LUNGCA study). J Natl Cancer Inst. 2025 Jul 1;117(7):1474-1484. doi: 10.1093/jnci/djaf061. PMID 40131728
- [Background] Xia L, Mei J, Kang R, Deng S, Chen Y, Yang Y, Feng G, Deng Y, Gan F, Lin Y, Pu Q, Ma L, Lin F, Yuan Y, Hu Y, Guo C, Liao H, Liu C, Zhu Y, Wang W, Liu Z, Xu Y, Li K, Li C, Li Q, He J, Chen W, Zhang X, Kou Y, Wang Y, Wu Z, Che G, Chen L, Liu L. Perioperative ctDNA-Based Molecular Residual Disease Detection for Non-Small Cell Lung Cancer: A Prospective Multicenter Cohort Study (LUNGCA-1). Clin Cancer Res. 2022 Aug 2;28(15):3308-3317. doi: 10.1158/1078-0432.CCR-21-3044. PMID 34844976